CLINICAL TRIAL: NCT04633824
Title: Health Disparities on the Labor Floor
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Patrick T Hussey, Principal Investigator, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300006294; UAB (Other: Anesthesiology)
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pain; Pregnancy Related
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with private insurance
  Interventions: Other: Retrospective Electronic Medical Record Review
- Patients with public/self-payer insurance
  Interventions: Other: Retrospective Electronic Medical Record Review

INTERVENTIONS:
Other: Retrospective Electronic Medical Record Review — Patients will be assessed retrospectively for evidence of successful or failed epidural extension in the setting of need for cesarean section

SUMMARY:
The Agency for Healthcare Research and Quality (AHRQ) defines a disparity as a difference or a gap that exist between two groups, which is both statistically significant, larger than 10%, and indicates poor quality for the minority (non-referent) group. Despite advances in public health initiatives and medicine, disparities in healthcare are persistent. For example, in the United States, maternal mortality ratio has doubled since 1987 to 2009 where African American women were 4 times as likely to die from childbirth. Although there was no observed racial disparity in maternal deaths at University of Alabama Birmingham, there is anecdotal experience that may suggest health disparities do exist on the labor floor when examining neuraxial utilization and effectiveness. This retrospective study will seek to examine the successful extension of labor analgesia for cesarean section as it relates to insurance status.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Age >/= age 18 years

Exclusion Criteria:

* Women less than age 18 will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women admitted to the labor and delivery unit from 1/1/2015 to 12/31/2019, who meet the above defined inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Successful extension of labor epidural catheter for cesarean section | from the time of admission to the time of delivery
  labor epidural activation in the setting of cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hussey, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No